CLINICAL TRIAL: NCT01357200
Title: Enteral Formula Tolerance in the Obese Critical Care Population
Brief Title: Feeding Trial in the Obese Critical Care Population
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 10.02.US.CLI
Record Dates: First submitted 2011-05-15; First posted 2011-05-20 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Critical Illness; Obesity
MeSH Terms: conditions — Critical Illness; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critically ill obese adults: Age ≥ 18 years, body mass index (BMI) ≥ 30, in intensive care unit (ICU) requiring tube feeding ≥ 3 days
  Interventions: Other: enteral formula

INTERVENTIONS:
Other: enteral formula — Complete feeding of study enteral formula, route and regime prescribed by the physician.

SUMMARY:
This study will assess enteral feeding in an obese critically ill population with a higher protein whey based peptide formula.

DETAILED DESCRIPTION:
Assess enteral feeding goal with a higher protein whey based peptide formula in an obese critically ill population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Surgical or Medical intensive care unit (ICU) patient
* Body mass index (BMI) ≥ 30

Exclusion Criteria:

* pregnant or lactating
* unable to access gastrointestinal (GI) tract for feeding via tube
* other contraindication to tube feeding
* admitted with burns
* severe head trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill obese adults
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
time to feeding goal achievement | up to 5 days
  on all participants

SECONDARY OUTCOMES:
gastrointestinal measures assessment | daily for up to 11 days
  on all participants
percent of nutrition goal met | up to 5 days
  on all participants
serum biochemical markers assessment | daily for up to 11 days
  on all participants
assessment of frequency and nature of adverse events | daily for up to 11 days
  on all participants

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky